CLINICAL TRIAL: NCT04660578
Title: A.Chohan Continuous Squeezing Suture (ACCSS) for Controlling Hemorrhage From the Lower Uterine Segment at the Cesarean Section for Placenta Previa / Accreta: a Case Series
Brief Title: A.Chohan Continuous Squeezing Suture (ACCSS) for Placenta Previa / Accreta
Acronym: ACCSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 497/RC/KEMU; SMDC/SMRC/97-19 (Other: Sharif Medical and Dental College, Lahore, Pakistan)
Record Dates: First submitted 2020-11-29; First posted 2020-12-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Placenta Previa With Hemorrhage - Delivered; Placenta Accreta
Keywords: Postpartum hemorrhage; Peripartum hysterectomy
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): A.Chohan continuous squeezing suture (ACCSS); An Obstetrical procedure using half circle 40mm round body polyglactin 910 suture #1 (Vicryl plus by Ethicon®), for controlling hemorrhage from the lower uterine segment, in patients with placenta previa / accreta for the prevention of hysterectomy at cesarean section.
  Interventions: Procedure: ACCSS

INTERVENTIONS:
Procedure: ACCSS — A. Chohan Continuous Squeezing Suture (ACCSS)

SUMMARY:
Placenta praevia and accreta spectrum disorders are rising in incidence due to increased rate of repeat caesarean sections. Peripartum hysterectomy remains the only definitive treatment of massive postpartum haemorrhage related to this condition. A multitude of conservative treatments is described in literature, which includes pelvic devascularization under radiological control, myometrial resection with placenta in situ, and various suturing techniques some involving inversion of cervix. Variable success rates are described, but search continues for a simple, safe and effective treatment. Such a surgical technique i.e. A. Chohan Continuous Squeezing Suture (ACCSS) is described in this study for controlling haemorrhage from the lower uterine segment at caesarean section for placenta praevia and accrete spectrum disorders.

DETAILED DESCRIPTION:
Postpartum haemorrhage (PPH) has always been a prominent cause of maternal morbidity as well as mortality worldwide, with uterine atony as the leading cause and peripartum hysterectomy as the only definitive treatment option . Researchers are struggling throughout the years to find a treatment modality other than hysterectomy, which has least morbidity and potential to preserve fertility. In an attempt to find a non-radical treatment for PPH due to uterine atony, a novel uterine compression suture was introduced in 1997. The time then witnessed emergence of a series of its variants from all over the world which effectively lowered the incidence of peripartum hysterectomy from uterine atony.

Meanwhile the incidence of placenta praevia and placenta accreta spectrum disorder rose dramatically across the globe because of rising incidence of repeat caesarean sections. Placenta accreta spectrum has opened up a new era in the history of PPH, as forcible separation of adherent placenta leads to massive bleeding from placental bed. Peripartum hysterectomy has once again emerged as gold standard treatment for this variety of PPH with its overall morbidity of 40-50%, and mortality of 7-10% in case of placenta percreta. The fear of placental bed bleeding has led to the development of conservative managements like "leaving the placenta in situ approach" with its wide range of mild to severe, and serious morbidities. The conservative surgical techniques i.e. The triple P procedure, one step conservative surgery approach, have also used the concept of non-separation of placenta and have instead adopted resection of myometrium with placenta in situ. These surgeries involve devascularisation of deep pelvic / major abdominal vessels and ligation of complex arterial anastomosis making the procedure technically difficult. Moreover, the devascularisation is done under extensive and expensive interventional radiological equipment which places the procedures out of reach for the routine setups particularly in the under developed countries. Another conservative surgical technique i.e. stepwise surgical approach, which described separation of placenta also mainly relied upon devascularisation of pelvic organs by bilateral ligation of anterior branch of internal iliac artery rather than elaborating the details of technique of controlling haemorrhage at the actual bleeding site.

Three corners stones of uterine compression sutures have been described in literature i.e. simplicity, safety and efficacy and no such suturing technique so far is published. Hence, it's the time for innovation in the treatment of placenta praevia and PAS. In this study, we report our own experience of a conservative surgical technique i.e. A. Chohan Continuous Squeezing Suture (ACCSS) application in the lower uterine segment during caesarean section in profusely bleeding patients with placenta praevia and placenta accreta spectrum without involvement of urinary bladder and other pelvic organs. This surgical technique takes on the separation of placenta and describes a placental bed suturing without involvement of interventional radiology as well as ligation of deep pelvic vessels. The objective of this study is to assess the simplicity, safety and efficacy of this surgical technique in the management of PAS, with the intension to develop a simple, safe and effective alternative to hysterectomy.

Surgical Procedure:

After opening the abdomen, a transverse incision was given in the lower uterine segment after ascertaining the site of easy fetal access avoiding the placenta as far as possible. After the delivery of the baby, the uterus was exteriorized and routine uterotonics were given. The placenta was left in-situ and incision margins were held with Green-armitage forceps to minimize bleeding.

The urinary bladder was dissected away to allow suturing on the inner side of the lower uterine segment. Uterine arteries were ligated on both sides and any blood vessels on the way were secured immediately. The placenta was then removed completely.

Within the puddle of blood, the ring of internal os was identified with the index and middle finger of one hand and held with Babcock forceps with the other hand. On the exposed inner surface of the LUS, suturing was started from the left corner of uterine incision, taking multiple half cm bites through half-thickness of the tissue at half cm intervals to reach the outer half of ring of the internal os. The suture was then tied and knot secured causing squeezing of uterine tissue. From here onwards similar sutures were placed continuously at 1 cm distance till the right corner was reached, where the knot was secured. During suturing it was ensured that internal os remains patent. The continued pull on the suture caused the squeezing of the LUS and arrested bleeding from all sinuses present at the placental site. If the bleeding was seen on the posterior uterine wall, a similar suture was applied. It was started from the outer half of the posterior lip of the ring of the internal os and going up to the highest bleeding point on the posterior wall of the uterus, extending from the left to right end of the uterine incision.

Any left over bleeding points were secured with separate hemostatic sutures, Routine closure of the uterus was performed in two layers as in the lower segment cesarean section.

The hospital stay of the patients was 3-7 days. All patients were reviewed on 7th postoperative day and were inquired about the history of fever, abdominal pain and excessive vaginal bleeding. The character of vaginal discharge / lochia was noted and any urinary complaint recorded. Caesarean section wound was examined and stitches removed. Second follow up visit was at 6 weeks postpartum for similar assessment and record of lactation / menstruation status. Pelvic ultrasound was done on both visits to detect any pelvic organ abnormality and collection of blood or pus.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting patients at 32 weeks of gestation, with the diagnosis of placenta previa and placenta accreta spectrum without involvement of bladder and other pelvic organs.
2. Woman who wished to conserve the uterus.

Exclusion Criteria:

1. Patients were excluded from the study if an emergency cesarean section was done due to severe antepartum hemorrhage before the plan of surgery.
2. Patients with Placenta accreta spectrum with bladder and/or other pelvic organ involvement.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Peripartum hysterectomy | 24 hours
  Number of peripartum hysterectomies within the study group

SECONDARY OUTCOMES:
Application time of suture in minutes | within 20 minutes
  Time taken by the surgeon to complete application of suture in minutes
Estimated blood loss | duration of surgery in minutes
  Estimate of blood loss in milliliters (ml) within the duration of cesarean section
Number of units of blood transfusions | First 24 hours
  number of units of blood transfused intra-operatively and within first 24 hours
Duration of stay of the participants in hospital in days | 7 days
  Number of days the patient stays in hospital postoperatively
Number of patients requiring other conservative medical and surgical treatments | Duration of surgery in minutes
  use of additional measures (oxytocin, tranexamic acid, prostaglandins, uterine packing, internal iliac artery ligation) to control intraoperative hemorrhage from the lower uterine segment
Number of patients with urinary bladder trauma and its complication | 6 weeks
  Intraoperative urinary bladder damage or any complication arising from it within 6 weeks of surgery
Number of patients with secondary postpartum hemorrhage | 6 weeks
  Hemorrhage in milliliters (ml) after 1st 24 hours and before 6 completed weeks of surgery
Prevalence of maternal mortality | 6 weeks
  Number of mothers dying in relation to cesarean section within 6 completed weeks of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Chohan, FRCOG, FCPS, Principal Investigator — King Edward Medical University, Lahore, Pakistan
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngwenya S. Postpartum hemorrhage: incidence, risk factors, and outcomes in a low-resource setting. Int J Womens Health. 2016 Nov 2;8:647-650. doi: 10.2147/IJWH.S119232. eCollection 2016. PMID 27843354
- [Background] Mousa HA, Blum J, Abou El Senoun G, Shakur H, Alfirevic Z. Treatment for primary postpartum haemorrhage. Cochrane Database Syst Rev. 2014 Feb 13;2014(2):CD003249. doi: 10.1002/14651858.CD003249.pub3. PMID 24523225
- [Background] Dohbit JS, Foumane P, Nkwabong E, Kamouko CO, Tochie JN, Otabela B, Mboudou E. Uterus preserving surgery versus hysterectomy in the treatment of refractory postpartum haemorrhage in two tertiary maternity units in Cameroon: a cohort analysis of perioperative outcomes. BMC Pregnancy Childbirth. 2017 May 30;17(1):158. doi: 10.1186/s12884-017-1346-0. PMID 28558661
- [Background] Yong S, Pradhan M. Intrauterine Gauze Packing in Primary Post Partum Hemorrhage following Caesarean section: A Clinical study. Nepal J Obstet Gynaecol. 2013;7(1):33-6.
- [Background] D D, Reginald P. Internal uterine tamponade. A Textb Postpartum Hemorrhage. 2006;263-7.
- [Background] B-Lynch C, Coker A, Lawal AH, Abu J, Cowen MJ. The B-Lynch surgical technique for the control of massive postpartum haemorrhage: an alternative to hysterectomy? Five cases reported. Br J Obstet Gynaecol. 1997 Mar;104(3):372-5. doi: 10.1111/j.1471-0528.1997.tb11471.x. PMID 9091019
- [Background] Selcuk I, Uzuner B, Boduc E, Baykus Y, Akar B, Gungor T. Step-by-step ligation of the internal iliac artery. J Turk Ger Gynecol Assoc. 2019 May 28;20(2):123-128. doi: 10.4274/jtgga.galenos.2018.2018.0124. Epub 2018 Nov 30. PMID 30499283
- [Background] Wang CY, Pan HH, Chang CC, Lin CK. Outcomes of hypogastric artery ligation and transcatheter uterine artery embolization in women with postpartum hemorrhage. Taiwan J Obstet Gynecol. 2019 Jan;58(1):72-76. doi: 10.1016/j.tjog.2018.11.014. PMID 30638485
- [Background] Lee HY, Shin JH, Kim J, Yoon HK, Ko GY, Won HS, Gwon DI, Kim JH, Cho KS, Sung KB. Primary postpartum hemorrhage: outcome of pelvic arterial embolization in 251 patients at a single institution. Radiology. 2012 Sep;264(3):903-9. doi: 10.1148/radiol.12111383. Epub 2012 Jul 24. PMID 22829685
- [Background] Matsubara S, Yano H, Ohkuchi A, Kuwata T, Usui R, Suzuki M. Uterine compression sutures for postpartum hemorrhage: an overview. Acta Obstet Gynecol Scand. 2013 Apr;92(4):378-85. doi: 10.1111/aogs.12077. Epub 2013 Feb 9. PMID 23330882